CLINICAL TRIAL: NCT00756860
Title: A Phase 1 Multiple Dose Study to Compare the Effects of AMG 223 and Sevelamer HCL (Renagel®) on Phosphate Binding in Healthy Volunteers
Brief Title: A Phase 1 Multiple Dose Study to Compare the Effects of AMG 223 and Sevelamer HCL (Renagel®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Organization: Amgen (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070885
Record Dates: First submitted 2008-09-11; First posted 2008-09-22 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sevelamer

ARMS (2):
- 2 (Active Comparator): 30 subjects will be randomized on Day -1
  Interventions: Drug: Renagel® (sevelamer hydrochloride)
- 1 (Experimental): 30 subjects will be randomized on Day -1
  Interventions: Drug: AMG 223

INTERVENTIONS:
Drug: AMG 223 — 2 g AMG 223 (4 x 500 mg capsules ) TID on Days 1 through 7
  Arms: 1
Drug: Renagel® (sevelamer hydrochloride) — 2g Renagel® (2 x 800 mg capsules + 1 x 400 mg capsule) TID on Days 1 through 7
  Arms: 2

SUMMARY:
The purpose of this study is to determine if subjects on 2g AMG 223 will achieve 60% or greater reduction in urinary phosphorus from baseline compared to subjects on 2g Renagel®.

Renagel®, Sevelamer HCl is currently the market leader for the treatment of hyperphosphatemia in patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking men and women between the ages of 18 and 45 years, inclusive the time of consent. Healthy is defined as an absence of clinically relevant abnormalities, as identified by a detailed medical history, complete physical examination, vital signs, 12 lead ECG, and clinical laboratory tests at Screening through randomization Females of child-bearing potential must be non-lactating, must have a negative serum pregnancy test before study enrollment, and must use a highly effective form of contraception for at least 3 months before study drug administration, during the study, and for an additional 1 month after study completion
* Male participants and/or their partners must use a highly effective form of contraception during sexual intercourse during the study and for an additional 1 month after study completion
* A body mass index (BMI) between 18 and 30 kg/m2, inclusive
* Serum phosphate within normal range
* Willing and able to provide written informed consent
* Willing and able to be confined to the clinical research unit (CRU) as required by the protocol
* Must abstain from any caffeine or alcohol within 72 hours of Day-7 through Day 7 inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant hematologic, renal, endocrinologic, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) judged to be relevant by the investigator
* History of bowel obstruction, dysphagia, swallowing disorders, gastrointestinal disorders such as inflammatory bowel disease, constipation, major gastrointestinal surgery, hemorrhoids, or gastric/duodenal ulcers
* Unable or unwilling to swallow numerous capsules/tablets
* Known hypersensitivity to Renagel® or its constituents
* Having an estimated glomerular filtration rate (GFR) < 80 ml/ min (Cockcroft Gault equation)
* Blood donation > 500 mL within 60 days of Screening
* History of alcohol abuse (more than 14 alcoholic drinks per week for men and 7 alcoholic drinks per week for women (one drink equals 12 oz beer, 8 oz of wine, or a drink containing one ounce of liquor) or use of illicit drugs within 12 months of Screening
* Positive results for the following tests:
* Urine drug and breath alcohol at Screening or Day -7,
* Serum pregnancy test (females only) at Screening or Day -7,
* Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HepCAb) at Screening
* Women who are pregnant, breastfeeding, or plan to become pregnant during the course of the study Participation in another clinical trial with any investigational drug or device within 30 days or 5 half lives of the investigational drug (if known), whichever is longer, of study drug administration
* Use of prescription and nonprescription drugs (herbal remedies, vitamins, and nutraceuticals) within 14 days or 5 half-lives, whichever is longer, before Day -7 and during the study (excluding acetaminophen at doses of 2 g/day and hormonal birth control pills)
* Use of prescription and nonprescription drugs that may affect gut motility within 14 days or 5 half-lives, whichever is longer, before Day -7 and during the study
* Subject will not be available for follow-up assessment or concerns for subject's compliance with the protocol procedures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the effects of 2g AMG 223 and 2g Renagel® on 24 hour urinary phosphorous excretion after multiple doses in healthy volunteers. | Including the 28-day Screening period, the 15-day residency period, and the follow-up on Day 15 (one week after discharge from the clinical research unit), the maximum subject participation is approximately 50 days.

SECONDARY OUTCOMES:
To compare the effects of 2g AMG 223 and 2g Renagel® on 24 hour fecal phosphorous excretion after multiple doses in healthy volunteers. | Including the 28-day Screening period, the 15-day residency period, and the follow-up on Day 15 (one week after discharge from the clinical research unit), the maximum subject participation is approximately 50 days.
To assess safety and tolerability of multiple doses of 2g AMG 223 in healthy volunteers. | Including the 28-day Screening period, the 15-day residency period, and the follow-up on Day 15 (one week after discharge from the clinical research unit), the maximum subject participation is approximately 50 days.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com